CLINICAL TRIAL: NCT05707923
Title: How Single-Word and Telegraphic Simplification Affects Language Processing and Word Learning in Young Children With Autism Spectrum Disorder
Brief Title: How Simplified Language Affects Comprehension and Learning in Young Autistic Children
Acronym: PALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Courtney E. Venker, Assistant Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4584124; R01DC020165 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-02-01 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: language; autism; intervention; processing; learning; early childhood; treatment; early intervention; telegraphic; language input; looking-while-listening; eye tracking; comprehension; neurodevelopmental disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Language; Autistic Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Utterance Type (Experimental): This study uses a within-participant experimental manipulation. All participants will be exposed to all utterance types (across trials).
  Interventions: Behavioral: Linguistic simplification

INTERVENTIONS:
Behavioral: Linguistic simplification — Children will participate in screen-based language processing and word learning tasks in which they hear utterances with different types and amounts of linguistic simplification (i.e., a within-group manipulation).

SUMMARY:
The long-term study goal is to experimentally evaluate the components (and likely active ingredients) of early language interventions for young children with ASD. The overall objective is to determine how single-word and telegraphic simplification affects real-time language processing and word learning in young children with ASD (relative to full, grammatical utterances). The proposed project will investigate three specific aims: 1) Determine how single-word and telegraphic simplification affects language processing. 2) Determine how single-word and telegraphic simplification affects word learning. 3) Evaluate child characteristics that may moderate the effects of linguistic simplification on language processing and word learning. Aim 1 will test the hypothesis that children with ASD will process full, grammatical utterances faster and more accurately than single-word or telegraphic utterances. Aim 2 will test the hypothesis that full, grammatical utterances will support word learning better than telegraphic or single-word utterances. Aim 3 will test the hypothesis that language and cognitive skills significantly moderate the effects of linguistic simplification on language processing and word learning in young children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Existing or suspected autism spectrum disorder, confirmed through ADOS-2
* English as primary language
* 1-4 years old

Exclusion Criteria:

* Known genetic condition (e.g., Down syndrome, fragile X)
* Cerebral palsy
* Acquired brain injury
* Uncorrected vision or hearing impairment

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Gaze location on Looking-While-Listening (LWL) tasks | Single assessment per task; total duration less than 10 minutes per task
  LWL involves a child looking at a screen with two images, one on each side of the screen, while being provided an auditory cue that includes the name of the target image. The primary outcome is a dichotomous variable indicating whether the child is fixated on the target image or the distracter image; gaze directed at neither image will be considered missing. It will be determined whether gaze is to the left or right image, using trained coders who are blind to target side. Gaze location will be observed every 33 ms from 300 ms after onset to 2000 ms after target word onset, for a total of 51 observations per trial. Analyses will focus on differences across trial types and child characteristics in the trajectory of gaze location over the course of the trial.

SECONDARY OUTCOMES:
Gaze location in Teaching Phase of Study 2b (Fast Mapping) | Single assessment; total duration less than 10 minutes
  A secondary outcome measure will be gaze location during the Teaching Phase of the Fast Mapping task (Study 2b). The variable is a dichotomous variable indicating whether the child is fixated on the novel image (only a single image is presented in each trial during the Teaching Phase) or not. It will be determined whether gaze is directed to the novel image, as our prior attempts to manually code single-object trials have not been successful. Only children who successfully calibrate and provide adequate automatic eye-tracking data in the Fast Mapping task will be included. Gaze location will be observed every 33 ms during the Teaching Trials. Analyses will focus on differences across trial types (single-word vs. full, grammatical teaching utterances).

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Dataset will include eye-gaze data, assessment scores, and transcriptions. De-identified analyzed data will be shared with other scientists for non-commercial research purposes in accordance with Michigan State University policy. Pending informed consent, de-identified data will be uploaded to the National Database for Autism Research, and transcripts will be shared with ASDBank. Scientific resources generated will be made available prior to publication if the work is different from our purposes. Following publication, resources will be made available to the broader scientific community on request. Findings and de-identified data will be shared through a variety of avenues, including scientific and clinical conferences, webinars, newsletters and scholarly manuscripts. Identifiable data may be shared if a family provides consent. All peer-reviewed manuscripts will be submitted to NIH's PubMed Central, to be made available at least 12 months after the official publication date.